CLINICAL TRIAL: NCT07200648
Title: Basic Income Guaranteed: Los Angeles Economic Assistance Pilot
Acronym: BIG:LEAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: The City of Los Angeles (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 849819
Record Dates: First submitted 2025-09-09; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Financial Wellbeing; Psychological Distress; Physical Functioning; Housing; Food Security; Income; Educational Attainment; Health; Well-being/Quality of Life; Employment; Family Dynamics; Stress
Keywords: guaranteed income; cash transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guaranteed income (Experimental): $1,000 of unconditional cash per month for 12 months
  Interventions: Other: Unconditional cash transfer
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Unconditional cash transfer — $1,000 unconditional cash transfer per month for 12 months
  Other Names: Guaranteed income; Basic income; Guaranteed basic income; Cash transfer
  Arms: Guaranteed income

SUMMARY:
The goal of this randomized controlled trial is to learn if receipt of a guaranteed income works to reduce financial hardship and improve quality of life. The main questions it aims to answer are:

1. How does GI affect participants' quality of life?
2. What is the relationship between GI and participants' subjective sense of self?
3. How does GI affect participants' income, and through what mechanisms?
4. How does the implementation of GI inform the existing safety net?

Participants will:

Receive an recurring unconditional cash transfer of $1,000 per month every month for 12 months OR receive no unconditional cash transfer Complete surveys at six month intervals during the course of the study Be invited to participate in in-depth interviews

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* Resident of Los Angeles, CA,
* At or below 100% of Federal Poverty Level
* Have been negatively impacted by COVID-19
* Have a dependent

Exclusion Criteria:

* less than 18 years of age
* not a resident of Los Angeles, CA
* Above 100% of Federal Poverty Level
* Not negatively impacted by COVID-19
* Do not have a dependent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8194 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Psychological distress (Kessler 10) | Prior to baseline and at 6 month intervals until 6 months post-treatment
  Each item is scored from one 'none of the time' to five 'all of the time'. Scores of the 10 items are then summed, yielding a minimum score of 10 and a maximum score of 50. Scores totaling less than 20 indicate that a person is likely to be mentally well; scores between 20-24 suggest a person is likely to have a mild mental health disorder; 25-29 are likely to indicate a moderate mental health disorder; and those scoring 30 or higher are likely to have a severe mental health disorder.
Financial Wellbeing (CFPB Financial Well-Being Scale) | Prior to baseline and at 6 month intervals until 6 months post-treatment
  The Consumer Financial Protection Bureau's Financial Wellbeing Scale is scored from 0 to 100, where higher scores indicate a greater sense of financial well-being.
Physical functioning (SF-36) | Prior to baseline and at 6 month intervals until 6 months post-treatment
  Each response is scored as 0 (Yes, limited a lot); 50 (Yes, limited a little); or 100 (No, not limited at all). Averages closer to 100 indicate better physical functioning while averages closer to 0 indicate worse physical functioning.
Food security | Prior to baseline and at 6 month intervals until 6 months post-treatment
  4 items to assess past four week food insecurity: 1) worry about not having enough food, 2) inability to eat preferred foods, 3) having to eat foods that they did not want to eat, and 4) eating less because there was not enough food. Items scored as "yes" (1) or "no" (0).
Household environmental instability (CHAOS) | Prior to baseline and at 6 month intervals until 6 months post-treatment
  The Confusion, Hubbub, and Order Scale (CHAOS) is a 15-item scale that assesses household environmental instability. Each item is scored from 1 to 4. Scores of the items are then summed, with scores ranging from 15 to 60. The higher the score, the higher the level of environmental chaos in the home.
Mattering (Mattering Index) | Prior to baseline and at 6 month intervals until 6 months post-treatment
  The Mattering Index is a 24-item self-reported scale to assess an individual's sense of significance within their community and the extent to which they feel valued and recognized by others. The scale measures 3 dimensions of mattering: awareness (how people believe others perceive them), importance (how people believe that others are emotionally invested in them), and reliance (how much individuals feel others can rely on them). Item scoring is from 1 (strongly disagree) to 5 (strongly agree). The awareness dimension accounts for 8 items, with total scores ranging from 8 to 40. The importance dimension accounts for 10 items, with total scores ranging from 10 to 50. The reliance dimension accounts for 6 items, with total scores ranging from 6 to 30. Higher total scores in each domain indicate a greater sense of mattering.
Housing security | Prior to baseline and at 6 month intervals until 6 months post-treatment
  Three items to assess 1) housing status (e.g., renter, homeowner, rent-to-own, etc.), 2) past 6 month evictions (yes/no), and 3) past 5 year mortgage default notices (number of times). Evictions and mortgage defaults are scored as "1" if the response is greater than zero, and "0" if the response is zero.
Hope (Adult Hope Scale) | Prior to baseline and at 6 month intervals until 6 months post-treatment
  The Adult Hope Scale is a 12-item self-reported scale that assesses one's ability to set goals ("agency" subscale; 4 items) and the confidence to pursue them ("pathways" subscale; 4 items). Item scoring is from 1 (definitely false) to 8 (definitely true) and there are 4 filler items that are not scored. Subscale scores range from 4 to 32; total scores range from 8 to 64. Higher scores indicate higher hope.

SECONDARY OUTCOMES:
Intimate partner violence (Composite Abuse Scale) | Prior to baseline and at 6 month intervals until 6 months post-treatment
  The Composite Abuse Scale (CAS R-SF) is a 15-item scale designed to capture a respondent's experience of intimate partner violence (IPV) with a particular emphasis on the frequency of experiences. Respondents are asked whether they have experienced any of the 15 IPV items (e.g., My partner(s) shook, pushed, grabbed, or threw me). If they respond yes, they are asked to indicate how often it happened in the past 12 months (e.g., Not in the past 12 months, Once, A few times, Monthly, Weekly, Daily/Almost Daily), scored as 0 to 5. Total scores, ranging from 0 to 75, are computed by calculating the mean frequency of all abuse items and multiplying this score by 15, where there are responses for at least 11 of the 15 items (~70%). Scores for the psychological abuse (range: 0 to 30), physical abuse (range: 0 to 25), and sexual abuse (range: 0 to 10) subscales are calculated in the same manner. Higher scores indicate increased severity of experiences of intimate partner violence.
Access to recreational opportunities for children | Prior to baseline and at 6 month intervals until 6 months post-treatment
  Parent-reported participation by their child in enrichment activities (yes/no). If yes, parent-reported type of enrichment activity in which the child participated.
Neighborhood safety | Prior to baseline and at 6 month intervals until 6 months post-treatment
  Subsections of the Neighborhood Environment for Children Rating Scale cover worries about victimization and interactions with neighbors. Each item rated on a scale from 1 to 10, with 1 being "mostly false" and 10 being "mostly true." The scale score was calculated by adding the score for each of the individual items and dividing that sum by the number of non-missing items for that individual. Scores ranged from 0 to 10, with higher scores on the interaction subsection indicating more positive neighborhood interaction, and higher scores on the victimization subsection indicating more worry about harm to property, self, and others in the neighborhood.

CONTACTS AND LOCATIONS:
Overall Officials: Stacia West, PhD, Principal Investigator — The University of Tennessee; Amy Castro, PhD, Principal Investigator — The University of Pennsylvania; Bo-Kyung Elizabeth Kim, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Community Investment for Families Department - City of Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://upenn.box.com/v/CGIR-Report-LA-CA-BIGLEAP